CLINICAL TRIAL: NCT01538888
Title: Effects Whole Body Vibration in Ergospirometrics Parameters, Strength And Quality of Life: A Randomised Controlled Trial
Brief Title: Effects Whole Body Vibration in Ergospirometrics Parameters and Quality of Life
Acronym: EWBVEPQL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maíra F Pessoa, graduate, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EQ1
Record Dates: First submitted 2012-02-09; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: WHOLE BODY VIBRATION; AGED; VO2; muscle strength

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WHOLE BODY VIBRATION (Experimental): SEARCH THE CARDIOPULMONARY EFFECTS IN WHOLE BODY VIBRATION IN HEALTH ELDERLY
  Interventions: Procedure: WHOLE BODY VIBRATION

INTERVENTIONS:
Procedure: WHOLE BODY VIBRATION — 03 MONTHS, TWICE PER WEEK
  Other Names: POWER PLATE, MODEL MY3

SUMMARY:
This study makes sure that the training of whole body vibration induces changes in ergospirometric parameters, in strength and influence in quality of life in healthy elderly. A case that is run like a vibration training combined, increasing strength and VO2.

DETAILED DESCRIPTION:
The search use the spirometric values after whole body vibration training and resistance training

ELIGIBILITY:
Inclusion Criteria:

* aged 60 to 74 years
* sedentary or irregularly active according to the IPAQ short form with no known diseases

Exclusion Criteria:

* smoking
* acute hernia
* thrombosis
* labyrinthitis
* diabetes
* hemodynamic instability
* obesity
* osteoporosis
* neuromuscular diseases
* pulmonary comorbidities
* heart disease
* electrocardiographic changes during exercise
* taking medications that affected bone metabolism or muscle and don't adapt to any of the protocols

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
VO2 | 03 MONTHS IN INTERVENTION
  change to maximal oxygen consumption (ml.kg.min)in ergospirometric test after 03 months training in vibrating platform twice per weeck.

SECONDARY OUTCOMES:
quality of life | 03 month
  outcome measure with the SF 36 shot form (Medical Outcomes Study 36 - Item short form health survey)after 03 months training in vibrating platform twice per weeck

CONTACTS AND LOCATIONS:
Overall Officials: Maíra F Pessoa, MS, Study Director — Universidade Federal de Pernambuco; Rafaela B Sá, MS, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil